CLINICAL TRIAL: NCT02344277
Title: Evaluation of Subcutaneous Implantable Cardiac Defibrillator in Brugada Patients
Acronym: S-ICD Brugada
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC14_0238
Record Dates: First submitted 2015-01-16; First posted 2015-01-22 (Estimated); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Brugada Syndrome; S-ICD System (Implantable Defibrillator)
Keywords: Subcutaneaous Implantable Cardiac Defibrillator; Brugada syndrome; Effectiveness; Safety
MeSH Terms: conditions — Brugada Syndrome | interventions — Defibrillators, Implantable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: S-ICD System (implantable defibrillator) — The subjects will be symptomatic or asymptomatic Brugada patients with Indication for ICD replacement. Patients should be follow first at 1 month and then every 6 months according to the recent ACC/AHA/HRS guidelines60, for a period of 5 years until remote monitoring became available for S-ICD.
  Visit to 4 week post-implantation: Vital status, Clinical assessment data: weight; height; blood pressure; NYHA class, Exercise test will be performed to control sensing vectors during exercise, Electrocardiogram, Current cardiac medication, Device interrogation, Device programming, Save to USB pen drive data + Printouts Adverse events, Life quality evaluation form. Visit every 6 months post-implantation to 5 years follow-up visit: Vital status, Clinical status (e.g.NYHA) , Electrocardiogram , Current cardiac medication, Device interrogation, Device programming, Save to USB pen drive data + Printouts Adverse events, Life quality evaluation form, Current status of S-ICD system.

SUMMARY:
Brugada syndrome is an inherited arrhythmia syndrome with an increased risk of syncope and sudden death resulting from episodes of polymorphic ventricular tachychardia and fibrillation. Currently, there is no medical therapy for the Brugada syndrome and the only treatment available is the implantation of an ICD. There is no discussion on the interest of the ICD implantation in secondary prevention and in patients who experienced syncope but the best therapeutic is more difficult to draw in asymptomatic patients. Recently we demonstrated that in asymptomatic patients with a spontaneous type 1 aspect of Brugada syndrome, (i) there was a significant risk of ventricular arrhythmia, (ii) the problem of inappropriate shocks can be solve with a good ICD programming and (iii) the problem of lead failure remains the main problem in this young population very active and represent the main limitation to larger indication of ICD implantation in this population with a very long life expectancy as these patients had a normal life expectancy except the risk of ventricular arrhythmia.

In this context the S-ICD System (Boston Scientific Inc.) which is an implantable defibrillator technology that treats ventricular tachyarrhythmias using a subcutaneous pulse generator and electrode system rather than a transvenous lead system, represents a very attractive opportunity as it gives the possibility to protect the patients of the risk of ventricular arrhythmia with no risk of lead failure. However, as this is a new technology and as Brugada syndrome patients are a very specific population (very active patients, specific and changing over time ECG aspect that is at risk of T wave over sensing and high risk of SVT), it seems important to evaluate the effectiveness and the safety of S-ICD in this specific context.

ELIGIBILITY:
Inclusion Criteria:

- Patient with type I Brugada syndrome eligible for implantation of an S-ICD system:

Symptomatic : (history of resuscitated sudden death, syncope) with an ECG showing an aspect of Brugada syndrome type I before or after pharmacological tests (ajmaline or flecainide test) according to the criteria of the consensus conference and after ECG validation by the Clinical Events Committee experts.

Asymptomatic: with an aspect of spontaneous type I Brugada syndrome after ECG validation by the Clinical Events Committee experts.

* Brugada syndrome patient with Indication for ICD replacement.
* No contra-indication for S-ICD implantation (anatomic or physiologic criteria) with particular attention to the validation of the ECG prescreening implantation. For this study at least 2 vectors must be suitable for S-ICD implantation.
* Patients whose age is 18 years or above, or of legal age to give informed consent specific to state and national law.
* Patients who are willing and capable of providing informed consent, participating in all testing associated with this clinical investigation at an approved clinical investigational center.

Exclusion Criteria:

* Incessant ventricular tachycardia (VT) and/or documented spontaneous, frequently recurring VT that is reliably terminated with anti-tachycardia pacing.
* Patients with unipolar pacemakers or implanted devices that revert to unipolar pacing.
* Presence of any severe medical condition such that the patient is not expected to survive for the planned study follow-up period.
* Minor, patient under trusteeship or under guardianship.
* Patients who currently participate in an investigational drug or device that clinically interferes with the S-ICD-Brugada registry study endpoints and results.
* Female of childbearing potential without adequate contraception at the time of the implantation.
* Inability to comply with the follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects selected for participation will be symptomatic or asymptomatic Brugada patients and, implanted or not with any ICD. Site investigators are responsible for screening. Subjects must meet all inclusion criteria. Subjects with any exclusion criteria will be excluded. The recruitment of the patients will be performed in a selected number of centers specifically involved in the management of patients affected by the Brugada syndrome in Europe and in which databases of patients are available.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2015-05-12 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-25 (Actual)

PRIMARY OUTCOMES:
appropriate number of shocks to the number of shocks recorded at 5 years after S-ICD implantation | 5 years
  The primary endpoint is the rate of successful appropriate shocks recorded at 5 years after S-ICD implantation in Brugada syndrome patients. In this population that will be a mix of symptomatic and asymptomatic patients, we anticipate a 1.5% per year event rate that will allow us to have a total of 15 patients receiving an appropriate shock at the end of the study.

SECONDARY OUTCOMES:
annual rate of inappropriate shocks | 5 years
  The secondary end point will be the annual rate of inappropriate shocks, the complications of S-ICD implantation and the complications during the follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent PROBST, Pr, Principal Investigator — Nantes University Hospital
Locations (22):
- Denmark (2):
  - Copenhagen University Hospital, Copenhagen
  - Gentofte University Hospital, Gentofte Municipality
- France (16):
  - Bordeaux University Hospital, Bordeaux
  - Brest University Hospital, Brest
  - Grenoble University Hospital, Grenoble
  - Lille University Hospital, Lille
  - Hospices Civils de Lyon, Lyon
  - AP-HM La Timone, Marseille
  - Montpellier University Hospital, Montpellier
  - Nancy University Hospital, Nancy
  - Nantes University Hospital, Nantes
  - AP-HP Hôpital BIchât, Paris
  - Paris University Hospital - La pitié-Salpétrière, Paris
  - Rennes University Hospital, Rennes
  - La Réunion University Hospital, Saint-Pierre
  - Strasbourg University Hospital, Strasbourg
  - Toulouse University Hospital, Toulouse
  - Tours University Hospital, Tours
- University Medical Centre Mannheim, Mannheim, Germany
- University of Turin, Turin, Italy
- Spain (2):
  - Hospital clinic de Barcelona, Barcelona
  - Hospital Puerta de Hierro, Majadahonda